CLINICAL TRIAL: NCT03849092
Title: Financial Incentive of Abstinence From Smoking as a Means of Recruiting Smokers With Low Socioeconomic Status to Smoking Cessation Programs in Municipalities
Brief Title: Smoking Cessation: Financial Incentives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Charlotta Pisinger, Consultant Senior researcher Ass Prof, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 119404
Record Dates: First submitted 2018-02-22; First posted 2019-02-21 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Financial incentive (Experimental): 3 municipalities will receive 120.000 DKK for financial incentives.
  Interventions: Behavioral: Financial incentives
- Campaigns (Experimental): 3 municipalities will receive 120.000 DKK for campaigns.
  Interventions: Behavioral: Campaigns
- Control (No Intervention): 6 "clean" control municipalities perform their smoking cessation activities as usual. They wont receive any financial resources. These muncipalities have not been randomly selected but have been matched (by number of smokers attending the smoking cessation groups in the municipality in 2017, the year before the intervention). 3 of them are Campaing Control group and 3 are Finacial Incentives Control group.

INTERVENTIONS:
Behavioral: Financial incentives — Cessation programs in municipalities will offer a financial incentive of 1200 DKK to smokers who achieve continuous abstinence from smoking when attending a group-based smoking cessation program. Aimed at smokers with low socioeconomic status but other smokers are also included.
  Arms: Financial incentive
Behavioral: Campaigns — Municipalities will design anti-smoking campaigns targeting smokers, recommending to use a municipal free group-based smoking cessation program. Aimed at smokers with low socioeconomic status but other smokers are also included.
  Arms: Campaigns

SUMMARY:
The aim of this intervention is to test if the investigator, by offering a financial incentive to smokers who abstinence from smoking, can:

1. recruit more smokers with low socioeconomic status to municipal smoking cessation programs
2. achieve higher abstinence rates at municipal smoking cessation programs among citizens with low economic status - Rather than by use of campaigns (=usual strategy) informing citizens about their options for support at municipal smoking cessation programs?

DETAILED DESCRIPTION:
For decades the prevalence of smokers has been declining. However, during the last four years the prevalence is stagnated. All municipalities are offering support to/ and during smoking cessation. Nevertheless, a lot of the municipalities find it very difficult to recruit smokers to their programs - in particular smokers with low socioeconomic status.

Hypothesis: It is assumed that more smokers with low socioeconomic status, which are otherwise very difficult to reach with smoking cessation offerings, will attend in municipal smoking cessation programs if they are offered a financial incentive. It is also assumed that smokers with low socioeconomic status, who have difficulty quitting smoking, will achieve higher smoking cessation rates if they are offered a financial incentive of abstinence from smoking. The target group of this study is therefore smokers with low socioeconomic status (SES).

The study involves 6 intervention municipalities (3 financial incentives municipalities and 3 campaign municipalities), and 6 control municipalities. The investigator conducts matched randomization at municipality level, and matches the municipalities on number of smokers recruited to smoking cessation programs in the previous year (2017).

All 6 intervention municipalities receive 102.000 DKK (16536,43 UDS) which must be used on their intervention. Beside the intervention everything goes on as usual in each municipality. Each municipality is its own control and the change will be analyzed after the intervention. The prevalence of smokers in each municipality is registered as usual by means of the Health Profiles, however not in this study!, which aim not is to measure the number of citizens quitting smoking unaided, but solely aim to focus on the municipals smoking cessation activities.

1. Intervention in the 3 financial incentives municipalities: the municipalities will make simple invitations and advertisements, showing that smokers can achieve a financial incentive of 1200 DKK if they abstinence from smoking.

   The period of a smoking cessation program is 7 weeks, and participants will receive a financial incentive as a gift voucher the 4 last meeting days, if validated abstinent from smoking.
2. Intervention in the 3 campaign municipalities: each municipality decides how the campaigns/advertisement should look/be like. The campaign should try to target smokers with low SES, recommending getting support during smoking cessation.
3. Control municipalities: 6 "clean" control municipalities perform their smoking cessation activities as usual and do not receive any financial resources. They do not know that they are control group in a trial.

The investigators measure validated recruitment- and abstinence rates 6 and 12 months after last session.

ELIGIBILITY:
Inclusion Criteria:smoker. -

Exclusion Criteria: non smoker, vaping of e-cigarettes (only)

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1934 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Recruitment | 12 months
  Can we by offering financial incentives or by running a stop-smoking campaign recruit more smokers to municipal smoking cessation programs?
Smoking cessation rates | 6 months and 12 months
  Can we by offering financial incentives or by running a stop-smoking campaign achieve higher smoking cessation rates at municipal smoking cessation programs?

SECONDARY OUTCOMES:
Recruitment of smokers with low socioeconomic status | 6 weeks, 6 months and 12 months after quit date
  Can we by offering financial incentives or by running a stop-smoking campaign recruit more smokers with low socioeconomic status to municipal smoking cessation programs
Smoking cessation rates among citizens with low economic status | 6 weeks, 6 months and 12 months after quit date
  Can we by offering financial incentives or by running a stop-smoking camaign achieve higher smoking cessation rates at municipal smoking cessation programs among citizens with low economic status?

CONTACTS AND LOCATIONS:
Overall Officials: Charlotta Pisinger, Professor, MD, PhD, MPH, Principal Investigator — Centre for Clinical Research and Prevention
Locations (1):
- Center for Clinical Research and Prevention, Frederiksberg, Denmark

REFERENCES:
- [Derived] Pisinger C, Toxvaerd CG, Rasmussen M. Are financial incentives more effective than health campaigns to quit smoking? A community-randomised smoking cessation trial in Denmark. Prev Med. 2022 Jan;154:106865. doi: 10.1016/j.ypmed.2021.106865. Epub 2021 Nov 3. PMID 34740676